CLINICAL TRIAL: NCT07341425
Title: A Study Protocol for a Randomized Controlled Study of Focused Acceptance and Commitment Therapy (FACT)
Brief Title: Focused Acceptance and Commitment Therapy (FACT) for Stress, Anxiety, and Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-145-25
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-11

CONDITIONS: Focused Acceptance and Commitment Therapy (FACT); Wailist
Keywords: FACT; Focused Acceptance and Commitment Therapy; Brief interventions

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant information material intentionally omits detailed information about the FACT intervention and the specific aims of, for instance, comparing immediate versus waitlist. Instead, participants are informed that there is currently insufficient evidence to determine whether it is more beneficial to begin treatment immediately or after a waiting period, with good reasons to believe in both scenarios. This intentional concealment is deemed necessary to prevent potential expectation biases that could arise from participants' awareness of whether they will begin treatment immediately or wait, and how this might influence their perceptions of the potential benefits and drawbacks of the timing of therapy initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Acceptance and Commitment Therapy (FACT) (Experimental): The intervention is focused on cultivating three fundamental skills in FACT: 1) Openness 2) Awareness, and 3) Engagement. Individuals characterized by inflexibility tend to suffer because they suppress, control, or avoid private experiences (lack in openness), they overidentify with past/future thinking (lack in awareness), and/or disconnection from their values (lack in engagement). Participants randomized to the FACT group will receive therapy corresponding to a maximum of five sessions of up to 50 minutes each with up to 250 minutes of contact (e.g., 5 sessions of 50 minutes or brief phone sessions), which will be delivered flexibly across the three-month intervention period. Both the number and duration of sessions may vary based on participant needs, provided that the total therapy time does not exceed 250 minutes.
  Interventions: Other: Focused Acceptance and Commitment Therapy
- Wailist (No Intervention): The waitlist group will receive FACT after four months.

INTERVENTIONS:
Other: Focused Acceptance and Commitment Therapy — Focused Acceptance and Commitment Therapy: This is a short-term treatment to alleviate symptoms of stress, anxiety, and depression.
  Arms: Focused Acceptance and Commitment Therapy (FACT)

SUMMARY:
This study is an interventional study examining the feasibility and acceptability of Focused Acceptance and Commitment Therapy (FACT) as a short-term intervention. Sixty participants will be randomized to either an intervention group (FACT; receiving a maximum of 250 min treatment) or a waitlist control group (receiving treatment after four months). Inclusion criteria are elevated symptoms of anxiety (GAD-7 ≥ 9), depression (PHQ-9 ≥ 10), and/or stress (PSS ≥ 14). Participants will complete self-report questionnaires at baseline, post-treatment, and at 1- and 3-month follow-ups. Additionally, brief session questionnaires will be completed before and after each session. Recruitment will take place through general practi-tioners in the Aarhus area.

DETAILED DESCRIPTION:
The present study seeks to evaluate the feasibility, acceptability, and preliminary efficacy of FACT as a short-term, delivered-as-needed intervention (up to 5 sessions) compared to a waitlist group (receiving treatment as usual (TAU) during the waiting period). Specifically, the project aims to assess the feasibility of implementing FACT within a primary mental health care setting, its acceptability to individuals experiencing heightened distress, its potential to alleviate distress and improve psychological flexibility, and to explore when these changes occur.

The hypotheses for this study are as follows:

* Hypothesis 1: FACT is feasible and acceptable for treating people with psychological distress.
* Hypothesis 2: FACT will be more effective in reducing symptoms of psychological distress than the waitlist-group.
* Hypothesis 3: Clients receiving FACT will report greater psychological flexibility, sense of agency, and self-efficacy compared to the waitlist-group.

ELIGIBILITY:
Inclusion Criteria:

(i) age ≥ 18 years, (ii) clinically relevant symptoms of distress ≥ 4 [53] and either symptoms of anxiety measured with the Generalized Anxiety Disorders (GAD ≥ 9 [54]) questionnaire and/or symptoms of depression with assessed with the Patient Health Questionnaire (PHQ-9 ≥ 10 [55]) and/or symptoms of stress measured with the Perceived Stress Scale (PSS ≥ 14), (iii) Danish language proficiency, (iv) ability and willingness to give informed consent, (v) no or stable antidepressant/antianxiety medication (i.e., same dosage for ≥ 6 weeks), (vi) access to either a smartphone, tablet, or computer with a video camera

Exclusion Criteria:

(i) currently receiving other psychotherapy or counseling for the same problem, (iii) a history of bipolar disorder, (ii) current or past psychotic disorder, (iv) substance abuse or dependence judged to require treatment, (v) suicide risk requiring immediate hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disitress | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group. Assessments are also measured at the beginning of each FACT session.
  The Distress Thermometer [DT] measures participants' perceived level of psychological distress on a scale from 0 (no distress) to 10 (extreme distress).
Depressive symptoms | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group. Assessments are also measured at the beginning of each FACT session.
  Patient Health Questionnaire-9 [PHQ-9] consists of nine items and is rated on a four-point Likert scale ranging from 0 (not at all) to 3 (nearly every day). Total scores range from 0 to 27, with higher scores indicating more severe depression
Anxiety | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group. Assessments are also measured at the beginning of each FACT session.
  General Anxiety Disorder-7 [GAD-7] consists of 7 items scored from 0 (not at all) to 3 (nearly every day) with scores ranging from 0 to 21. Higher scores reflect more severe anxiety symptoms.
Stress | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group. Assessments are also measured at the beginning of each FACT session.
  Perceived Stress Scale-10 [PSS-10]. The scale consists of ten items rated from 0 (never) to 4 (very often), producing a total score between 0 and 40. Higher scores reflect greater levels of perceived stress.

SECONDARY OUTCOMES:
Valuing Questionnaire | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments were conducted at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group.
  Valuing Questionnaire [VQ] consists of ten items rated on a seven-point Likert scale from 0 (not at all) to 6 (completely true). The measure yields two subscales: Progress and Obstruction.
  * Progress (items, 3, 4, 5, 7,9. Range = 0 to 30) defined as enactment and perseverance in living consistently with one's values. Higher scores represent a closer alignment between one's internal values and one's actions.
  * Obstruction (items 1, 2, 6, 8, 10. Range = 0 to 30) represents the extent to which various disruptions got in the way of valued living. Higher scores represent more interference with living consistently with one's values.
Experiential avoidance | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group.
  The Brief Experiential Avoidance Questionnaire [BEAQ] consists of 15 items rated on a six-point Likert scale from 1 (strongly agree) to 6 (strongly disagree), yielding total scores between 15 and 90. Higher scores reflect greater levels of experiential avoidance.
Distancing from thoughts | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group.
  The Experience Questionnaire [EQ] includes 11 items on the decentering scale, each rated on a 5-point Likert scale from 1 (never) to 5 (all the time). Scores on the 11 items are summed to produce a total scale score, which can range from 11 to 55, with higher scores indicating greater levels of decentering.
Sense of Agency | Assessed at baseline; 3-months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8, and 10 months for the waitlist group.
  The Sense of Agency Scale [SoA] consisting of 13 items with responses recorded on a scale from 1 (strongly disagree) to 7 (strongly agreee). It measures Sense of Positive Agency (SoPA) and Sense of Negative Agency (SoNA). SoPA refers to a person's experience of having control over their body, thoughts, and environment. SoNA, in contrast, describes the experience of feeling that these aspects are not under one's control.
Self-compassion | Assesed at baseline; 3 months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8 and 10 months for the waitlist group.
  The Self Compassion Scale - short revised [SCS - SF] is rated on a five-point Likert scale (1 = almost never, 5 = almost always), with higher total scores indicating higher self-compassion.
Trust in the system | Assesed at baseline; 3 months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8 and 10 months for the waitlist group.
  The Health Confidence Score [HCS] s rated on a four-point Likert scale. For analysis, response options are scored from 0 to 3, with 'strongly agree' = 3, 'agree' = 2, 'neutral' = 1, and 'disagree' = 0. Higher scores indicate greater health confidence.
Use of Health Services | For the FACT group, assessments will be conducted post-treatment at 3 months and at follow-up at 4 months. For the waitlist group, assessments will be conducted at 3, 4, 7, and 8 months.
  Participants will be asked to report whether they receive any (additional) treatment related to the present-ing issue for which they initially sought help, and if so, the type and number of visits during the interim pe-riod. Reported treatments will be categorized into four types of health services: (1) Psychological services (e.g., sessions with a psychologist or psychotherapist); (2) Medical services (e.g., consultations with a psy-chiatrist, including pharmacological treatment); (3) Alternative treatments (e.g., reflexology, craniosacral therapy); and (4) Physical health services (e.g., physiotherapy or chiropractic care).
Physical activity | Assesed at baseline; 3 months post-intervention; follow-up at 4 months. Additional assessments at 6 months for the FACT group and at 7, 8 and 10 months for the waitlist group.
  Number of minutes spent on physical activity involving strength training, ball games or activities that raise your heart rate in the past week.
Session duration | Assessed at every FACT session
  At each FACT session, the duration of time spent in-session will be recorded.

OTHER OUTCOMES:
Working alliance | This questionnaire is only evaluated at the end of the first session
  Working Alliance Inventory - Short Revised [WAI-SR] consists of 12 items, each rated on a 5-point Likert scale from 1 (seldom) to 5 (always). Total scores range from 12 to 60, with higher scores indicating a stronger therapeutic alliance
Harm | This questionnaire is administered only post-treatment: at 3 months for the FACT group and at 7 months for the waitlist group.
  The Negative Effects Questionnaire [NEQ] consists of 20 items and is a self-report measure comprising three parts. First, respondents indicate whether each negative effect occurred during treatment using a yes/no format (coded as 1/0). Second, they rate the severity of each endorsed negative effect on a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), with higher scores reflecting greater severity. Third, respondents attribute each negative effect either to "the treatment I received" (coded as 1) or to "other circumstances" (coded as 0).
Feasibility: within-group effect | Will happen after the therapy has ended.
  The following feasibility criteria will be evaluated: 1) within-group effect of Cohen's d >.5,
Fidelity to the intervention | Will happen after the therapy has ended.
  Fidelity of the interventions. Fidelity assessment of session recordings will include two components: 1) adherence to key FACT principles (i.e., whether the key therapeutic elements were delivered as intended) and 2) therapist competency, with both aspects rated on a 0-2 scale. Two independent raters will evaluate a random sample of 20% of cases in the FACT group, covering all sessions for each selected participant.
Minimal harm | This questionnaire is administered only post-treatment, at 3 months for the FACT group and at 7 months for the waitlist group.
  Minimal harm evaluated with NEQ
Propective acceptability | CEQ will be measured at post session one.
  Prospective acceptability: Credibility/Expectancy Questionnaire for evaluating expected improvement of therapy [CEQ] will be measured post session one.
Retrospective acceptability | CSQ-8 will be measured at post treatment: 3 months for the FACT group and 7 months for the waitlist group.
  Retrospective acceptability: Client Satisfaction Questionnaire [CSQ-8], interest and usefulness of intervention [73].